CLINICAL TRIAL: NCT06902025
Title: An Early Exploratory Clinical Study on the Safety, Tolerability, and Preliminary Efficacy of JY231 Injection in the Treatment of Relapsed or Refractory B-cell Acute Lymphoblastic Leukemia (B-ALL)
Brief Title: JY231(JY231) Injection for the Treatment of Relapsed or Refractory B-Cell Leukemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: He Huang (Other)
Responsible Party: Sponsor-Investigator, He Huang, Professor, Director of the Bone Marrow Transplantation Center, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JY-CT-24-008
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: B-ALL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single-center, open, single arm study (Experimental): JY231 Injection for the treatment of relapsed or refractory B-cell Acute Lymphoblastic Leukemia (B-ALL) subjects who meet the inclusion criteria will receive a single intravenous injection of JY231, followed by regular observation and follow-up of the subject.
  Interventions: Drug: JY231 Injection

INTERVENTIONS:
Drug: JY231 Injection — Patients were enrolled and given a single dose of JY231 injection intravenously, hospitalized for observation over the following month, and followed up for observation over the following 15 years.

SUMMARY:
This study is an investigator-initiated single center, single arm clinical study with a target population of patients with relapsed or refractory B cell leukemia. It is an early exploratory clinical study of the safety, tolerability and initial efficacy of JY231 injection in the treatment of relapsed or refractory B-cell Acute Lymphoblastic Leukemia (B-ALL).

DETAILED DESCRIPTION:
This is an open-label, single-arm study to evaluate the efficacy and safety of in vivo Chimeric Antigen Receptor T-Cell(CAR-T cell) therapy in patients with relapsed refractory B-cell Acute Lymphoblastic Leukemia (B-ALL). Upon enrollment, subjects will receive an intravenous infusion of the JY231 preparation. Following the infusion, subjects will be hospitalized for one month for observation, and subjects will be evaluated for safety and efficacy. Subjects will be followed for up to 15 years to determine if the disease is under control.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~75 years old, gender is not limited;
2. Patients with a diagnosis of Cluster of Differentiation 19 positive(CD19+) B-ALL confirmed by flow cytometry or immunohistochemistry according to the criteria of the National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines for Acute Lymphoblastic Leukemia (2016.v1);
3. Meet the diagnosis of relapsed/refractory (relapsed/refractory) r/r CD19+ B-ALL, including any of the following:

   A.relapse within 12 months of first remission; B.initial refractory treatment that does not achieve complete remission after two doses of standard chemotherapy, or complete remission or relapse after first-line or multiple lines of salvage therapy;

   C.Patients with Ph+-ALL (Philadelphia chromosome-positive) in whom relapse or refractory is defined as meeting any of the following:

   ① Relapse or refractory after treatment with at least two tyrosine kinase inhibitor (TKI) agents or intolerance to TKI-type agents;

   ② Resistance or failure to achieve remission after receiving second-line TKI therapy;

   ③ Not suitable for TKI therapy;
4. Bone marrow cytomorphology with >5% prolymphocytes + juvenile lymphocytes; or flow Minimal Residual Disease(MRD) >=0.01%
5. Serum total bilirubin ≤ 51 mol/L, serum alanine aminotransferase (ALT) and azelaic transaminase (AST) both ≤ 3 times the upper limit of the normal range, blood creatinine ≤ 176.8 mol/L, and platelets ≥ 20×109/L;
6. Echocardiography showed left ventricular ejection fraction (LVEF) ≥50%;
7. Subjects without active pulmonary infection and inspiratory finger pulse oxygen saturation ≥92%;
8. Subjects have not received radiotherapy, chemotherapy, monotherapy or other anti-ALL therapy within 1 week prior to screening;
9. Predicted survival of 3 months or more;
10. Eastern Cooperative Oncology Group(ECOG) score of 0-2;
11. Subjects or their legal guardians volunteered to participate in this study and signed an informed consent form;

Exclusion Criteria:

1. Subjects with active central nervous system (CNS) leukemia;
2. Subjects with a history of active CNS disease such as seizures, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement;
3. Subjects who have been treated with another investigational drug within 30 days prior to screening or are still in the washout period;
4. Subjects who have had radiation therapy within 2 weeks prior to infusion;
5. Subjects with uncontrolled acute life-threatening bacterial, viral, or fungal infections (e.g., positive blood cultures ≤ 72 hours prior to infusion);
6. Subjects with unstable angina and/or myocardial infarction within 6 months prior to Screening;
7. Subjects with other prior or concurrent malignancies, with the following exceptions:

   ① Adequately treated basal cell, papillary thyroid, or squamous cell carcinoma (adequate wound healing is required prior to enrollment in the study);

   ② Cancer in situ of the cervix or breast that has been curatively treated and shows no signs of recurrence for at least 3 years prior to study entry;

   ③ primary malignancy that has been completely resected and in complete remission for ≥ 5 years.
8. Presence of subjects with arrhythmias not controlled by medical management;
9. Subjects with active neurologic autoimmune or inflammatory conditions (e.g. Guillain-Barre syndrome, amyotrophic lateral sclerosis);
10. Women who are pregnant or breastfeeding, and female subjects who plan to become pregnant within 2 years of their JY231 injection infusion or male subjects whose partners plan to become pregnant within 2 years of their JY231 injection infusion;
11. Subjects who, in the investigator's judgment and/or clinical criteria, have a contraindication to any of the investigational procedures or have other medical conditions that may place them at unacceptable risk.
12. Other conditions that, in the opinion of the investigator, should not be enrolled in this clinical study, such as poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events(AE) after infusion | Day 28、Month 2、Month 3、Month 6、Month 12、Month 18、Month 24
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included.
Maximal Tolerated Dose(MTD) | Up to 28 days after infusion
  MTD will be determined based on Dose-Limiting Toxicity(DLTs) observed during the first 28 days of study treatment.

SECONDARY OUTCOMES:
Objective Response Rate | Day 28、Month 2、Month 3、Month 6、Month 12、Month 18、Month 24
  Objective Response Rate(ORR) is defined as the proportion of subjects achieving complete remission(CR) and partial response(PR).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No